CLINICAL TRIAL: NCT01286896
Title: Use of Individual PK-guided Sunitinib Dosing: A Feasibility Study in Patients With Advanced Solid Tumors
Brief Title: Use of Individual Pharmacokinetically (PK)-Guided Sunitinib Dosing: A Feasibility Study in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M10PKS; 2010-021454-20 (EudraCT Number)
Record Dates: First submitted 2011-01-14; First posted 2011-01-31 (Estimated); Last update posted 2025-07-10 (Actual); Status verified 2011-10

CONDITIONS: Malignant Solid Tumour
Keywords: advanced solid tumors
MeSH Terms: interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sunitinib (Experimental): Sunitinib is administered in oral capsules of 12.5 mg. Patients will start with a continuous once-daily dose of 37.5 mg.
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Sunitinib — Patients will start treatment with a continuous once-daily dose of 37.5 mg sunitinib. After 22 days the first dose modification will be performed based on the total trough levels (TTL) combined for sunitinib plus SU12662 as measured by dried blood spot (DBS) analyses taken at day 15 ± 1day. A second dose modification will be performed after 36 days (7 days after the first dose adjustment) based on the TTL taken at day 29 ± 1day. One treatment cycle is defined as 28 days.
  After 8 weeks a third analyses for TTL will be performed without further consequences for sunitinib dosing. Patients will be evaluated by CT- or MRI-scans for the response to therapy at week 8, and thereafter every 12 weeks. One blood sample will be harvested for pharmacogenetic analyses.
  Other Names: Sutent®; SU 11248

SUMMARY:
The purpose of this prospective study is to determine the safety and feasibility of pharmacokinetically (PK) guided dosing of sunitinib in 30 patients.

At day 15 ± 1day, day 29 ± 1day and after 8 weeks ± 1day of sunitinib treatment sunitinib and SU12662 trough levels will be measured. Depending on the sunitinib and SU12662 trough levels (and toxicity) dose adjustments will be made.

DETAILED DESCRIPTION:
Sunitinib is an orally available inhibitor of vascular endothelial growth factor (VEGFR), platelet-derived growth factor (PDGF), cytokine receptor (c-KIT), and receptor tyrosine kinase (FLT-3) activity. Sunitinib is proven effective as single agent in several solid tumor types and is approved for use in advanced renal cell cancer (RCC) and imatinib-resistant or -intolerant gastrointestinal stromal tumors (GISTs). However, in a large percentage of patients (30 and 50%), dose reductions are required because of multiple grade 2 toxicities or due to grade 3 or 4 toxicities. Therefore, the currently used dosing schedule is not optimal.

Recently, a dose-efficacy relation was established for sunitinib treatment. This large meta-analysis of pharmacokinetic/pharmacodynamic data from studies performed in mRCC patients, GIST patients and patients with solid tumors, clearly showed a relationship between sunitinib exposure and efficacy and tolerability. Both time to progression (TTP) and overall survival (OS) were significantly better for mRCC patients with high area under the curve (AUC) compared to low AUC. This was not only observed for sunitinib exposure but also for its active metabolite SU12662. In addition, there was a significant relationship between exposure and probability of partial response (PR) or complete response (CR) in mRCC patients (p=0.00001), indicating that a dose intensity in patients should be as high as possible. Target plasma concentrations of sunitinib plus metabolite (N-desethyl sunitinib) are in the range of 50 to 100 ng/mL, as deduced from pharmacokinetic (PK) / pharmacodynamic (PD) preclinical data. Since the dose-efficacy relation for sunitinib treatment is solely established in a retrospective (meta-) analysis from patients treated in several studies, we propose to perform a prospective feasibility study in 30 patients with PK guided dosing of sunitinib. If PK guided once-daily continuous sunitinib dosing is feasible, a RCT in mRCC patients will be performed comparing PK guided dosing with a standard sunitinib dosing schedule.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically confirmed advanced tumors for which sunitinib is considered standard or patients with advanced or metastatic tumors for whom no standard therapy is available;
2. Age more then 18 years;
3. Able and willing to give written informed consent;
4. Able and willing to undergo blood sampling for pharmacogenetic and pharmacokinetic analysis;
5. Able and willing to undergo a tumor biopsy for DNA sequencing;
6. Able to swallow oral medications
7. Life expectancy more then 3 months, allowing adequate follow up of toxicity evaluation and antitumor activity;
8. WHO performance status of 0 or 1;
9. Evaluable disease according to RECIST 1.1 criteria;
10. Minimal acceptable safety laboratory values

    * ANC of => 1.5 x 109 /L
    * Platelet count of => 100 x 109 /L
    * Hepatic function as defined by serum bilirubin => 1.5 x ULN, ASAT and ALAT
    * 2.5 x ULN
    * Renal function as defined by serum creatinine => 1.5 x ULN or creatinine clearance => 50 mL/min (by Cockcroft-Gault formula);
11. No radio- or chemotherapy or other investigational drug treatment within the last 4 weeks prior to study entry, with the exception of palliative radiotherapy (8 Gy or on the extremities).

Exclusion Criteria:

1. Current treatment in another therapeutic clinical trial
2. Congestive heart failure, myocardial infarction or coronary artery bypass graft in the previous six months, ongoing severe or unstable angina or any unstable arrhythmia requiring medication
3. Patients with known alcoholism, drug addiction and/or psychotic disorders in the history that are not suitable for adequate follow up
4. Women who are pregnant or breast feeding.
5. Both men and women enrolled in this trial must agree to use a reliable contraceptive method throughout the study (definition of adequate contraceptive methods will be based on the judgment of the principal investigator or a designated associate).
6. Legal incapacity
7. Known allergy/intolerance to sunitinib or any of the excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2011-04-11 (Actual); Primary Completion 2011-12-27 (Actual); Study Completion 2011-12-27 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | During treatment with sunitinib Adverse Events will be recorded up to 30 days after treatment. Patient will remain on treatment untill the disease progression, 1 year in average
  To determine the safety and feasibility of PK guided dosing of sunitinib, weekly physical examination, blood hematology and blood chemistry parameters in the first 2 cycles, and monthly thereafter, will guide the safety of the treatment.

SECONDARY OUTCOMES:
objective response rate | 8 weeks after initiation and thereafter every 12 weeks until disease progression, 1 year in average
  To determine the objective response rate, CT-scan and/or MRI-scans will be performed 8 weeks after initiation of therapy and thereafter every 12 weeks until documented disease progression according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
time to tumor progression | Until the disease progression, 1 year in average
  To determine the time from start of study treatment to first documentation of objective tumor progression defined by 1.1 RECIST criteria performing CT/MRI scans 8 weeks after initiation of therapy and thereafter every 12 weeks
validating the associations between genetic markers | C1 D15 and C1 D29 and after 8 weeks
  To start with the validation of previously identified associations between genetic markers in the pharmacokinetic and pharmacodynamic pathways of sunitinib and the development of toxicities. At day 15 ± 1day, day 29 ± 1day and after 8 weeks ± 1day - PK: Fingerprick for dried blood spot analysis of total trough levels of sunitinib and SU12662.
  Once during cycle 1: EDTA blood samples for pharmacogenetic analyses
tumor biopsy and peripheral blood sample for DNA sequencing | Day -7
  Seven days prior to study medication treatment the tumor boipsy and blood draw will be performed to support the validation of DNA sequencing of tissue derived from a tumor biopsy and to obtain the DNA profile of the patient's tumor in order to (i) identify correlations between the genetic profile of the tumor and toxicity and efficacy parameters of sunitinib , and (ii) identify patients who could have advantage of specific follow-up treatment strategies.
Progression free survival | Untill disease progression, 1 year in average
  Measuring the time between the study start and the RECIST defined disease progression on CT/MRI scans performed 8 weeks after initiation of therapy and thereafter every 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Neeltje Steeghs, Md, PhD, Principal Investigator — The Netherlands Cancer Institute
Locations (1):
- The Netherlands Cancer Institute - Antoni van Leeuwenhoek Hospital, Amsterdam, Netherlands